CLINICAL TRIAL: NCT04640948
Title: High Flow Nasal Cannula Therapy for Initial Oxygen Administration in Acute Hypercapnic Respiratory Failure - A Comparison Study of Two Current Standards of Care
Brief Title: High VS Low Flow Nasal O2 for Acute Hypercapnic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19106MA-AS
Record Dates: First submitted 2020-09-11; First posted 2020-11-23 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Acute Hypercapnic Respiratory Failure; Acute Exacerbation of COPD
Keywords: Acute exacerbation of COPD; High flow nasal oxygen; High flow nasal insufflation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel group trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, the participants , care provider and investigator cannot be blinded but the outcome is objective and data will be analyzed by statistician independent of the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High flow nasal therapy (HFNT) (Experimental): Characterized by an elevated arterial CO2 (PaCO2) level of > 6kPa due to ventilatory failure. The ventilatory failure relates to the imbalance between the respiratory demand and the capacity of the respiratory system to match the demand.
  Interventions: Device: High flow nasal therapy
- Low flow oxygen (LFO) (Active Comparator): Characterized by an elevated arterial CO2 (PaCO2) level of > 6kPa due to ventilatory failure. The ventilatory failure relates to the imbalance between the respiratory demand and the capacity of the respiratory system to match the demand.
  Interventions: Device: Low flow oxygen

INTERVENTIONS:
Device: High flow nasal therapy — Controlled oxygen administration using at least 20 L/min of flow rate and titrated up as tolerated. Titration of supplemental oxygen to an arterial saturation between 88 - 92%.
  Other Names: High flow nasal insufflation
  Arms: High flow nasal therapy (HFNT)
Device: Low flow oxygen — Controlled oxygen administration using (venturi mask or nasal cannulae) titrated to an arterial saturation between 88 - 92% as the initial oxygen administration method with a flow rate of <20 L/min.
  Arms: Low flow oxygen (LFO)

SUMMARY:
Chronic lung conditions such as smoking related lung damage lead to breathing fail. This results in accumulation of gases such as carbon-di-oxide in the body especially during periods of illness known as exacerbation.

Current management of carbon-di-oxide accumulation is administration of oxygen, nebulisers, antibiotics etc and if necessary, provide a tight fitting mask around the face to provide breathing support. If this fails, then a patient is placed on a mechanical ventilator. The tight fitting mask therapy is also called non-invasive ventilation and is used widely but patients acceptability of the therapy is limited.

Providing a high flow of air with some oxygen could potentially provide the same benefit of the non-invasive ventilation and may also be better accepted by patients.

Currently the knowledge and evidence from studies suggest a beneficial role for this high flow therapy but this has not been investigated in well designed studies.

In the proposed study we aim to investigate whether use of the high flow therapy reduces the need for non-invasive ventilation in patients who present with a recent onset accumulation of carbon-di-oxide in their body due to long-term lung disease. If this shows benefit, it will lead to a bigger trial with patient benefiting by reduction in the non-invasive ventilation or indeed a need for an invasive breathing machine.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients > 18 years of age
2. Acute Hypercapnic respiratory failure with pH < 7.35 and pCO2 > 6 KPa

Exclusion Criteria:

1. Age < 18 years
2. Pregnant or Breast-Feeding
3. Patient cannot read and understand English
4. Hypercapnia secondary to a drug toxicity or non-pulmonary aetiology
5. Hypercapnia secondary to exacerbation of asthma
6. Contraindication to NIV
7. Contraindication to HFNC
8. Not for escalation to NIV
9. pH < 7.15
10. GCS 8 or less
11. Shock defined as systolic < 90 mmHg or a reduction by 20mmHg from usual systolic BP despite volume resuscitation
12. Respiratory or cardio-respiratory arrest
13. Any other indication that requires immediate invasive/non-invasive mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-06-13 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring NIV in each cohort | 6 hours
  Proportion of patients who require NIV by 6 hours of intervention.

SECONDARY OUTCOMES:
PaCO2 in Kilopascal | 1 hour, 6 hours and 24 hours.
  Blood arterial PCO2 level measured at the pre-specified timepoints or at the nearest timepoint.
PaO2 in Kilopascal | 1 hour, 6 hours and 24 hours.
  Blood arterial PaO2 level measured at the pre-specified time-points or at the nearest time-point.
pH | 1 hour, 6 hours and 24 hours.
  pH measured for acid-base status.
Respiratory rate (Breath/minute) | At 1 hour, 6 hours and 24 hours.
  Rate of breathing per minute as documented in medical notes.
Heart rate (Beat/minute) | 1 hour, 6 hours and 24 hours.
  Heart rate per minute as documented in medical notes.
Mean arterial pressure in millimeters of mercury | 1 hour, 6 hours and 24 hours.
  Mean arterial pressure in millimeters of mercury as documented in medical notes
Intubation rate | 1 hour, 6 hours and 24 hours.
ICU admission | From the date of randomization until the date of first documented admission to ICU, assessed up to 12 weeks.
In-hospital mortality | From the date of randomization until the date of death or hospital discharge, whichever came first, assessed up to 12 weeks.
ICU length of stay | From the date of ICU admission until the date of last documented ICU discharge or date of death from any cause, whichever came first, assessed up to 12 weeks.
Hospital length of stay | From the date of randomization until hospital discharge or date of death from any cause, whichever came first, assessed up to 12 weeks.
Dyspnoea | 1 hour, 6 hours and 24 hours.
  Dyspnoea will be assessed assessment using a visual analogue scale (VAS), score range 0-10, higher values represent a better outcome)) if patient has capacity or the Likert scale (score range 1-5; higher values represent a better outcome) to be completed by the clinical team (doctor/nurse/physio) if the patient lacks capacity.
Patient comfort | 1 hour.
  Comfort will be assessed assessment using a visual analogue scale (VAS), score range 0-10, higher values represent a better outcome)) if patient has capacity or the Likert scale (score range 1-5; higher values represent a better outcome) to be completed by the clinical team (doctor/nurse/physio) if the patient lacks capacity.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Mater Hospital, Belfast
  - Royal Victoria Hospital, Belfast

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared on request to the Principal Investigator and will be decided on a case by case basis.

REFERENCES:
- [Derived] Alnajada A, Blackwood B, Mobrad A, Akhtar A, Shyamsundar M. High-flow nasal cannula therapy for initial oxygen administration in acute hypercapnic respiratory failure: study protocol of randomised controlled unblinded trial. BMJ Open Respir Res. 2021 Jan;8(1):e000853. doi: 10.1136/bmjresp-2020-000853. PMID 33419742